CLINICAL TRIAL: NCT01264380
Title: A Phase I, Randomized, Open-label, Multi-center, Two Period Crossover Study to Investigate the Effect of Food on the Pharmacokinetics of a Single Oral Dose of RO5185426, Followed by Administration of 960 mg RO5185426 Twice Daily to BRAF V600E Positive Metastatic Melanoma Patients
Brief Title: A Study of the Effect of Food on the Pharmacokinetics of Single Dose RO5185426 And the Safety And Efficacy of Continuous Administration in Patients With BRAF V600E Mutation-Positive Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP25396
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: RO5185426
- 2 (Experimental)
  Interventions: Drug: RO5185426
- C (Experimental)
  Interventions: Drug: RO5185426

INTERVENTIONS:
Drug: RO5185426 — Single oral dose, fasted
  Arms: 1
Drug: RO5185426 — Single oral dose, with high fat meal
  Arms: 2
Drug: RO5185426 — Continuous administration, orally twice daily
  Arms: C

SUMMARY:
This randomized, open-label, two period crossover study will evaluate the effect of food on the pharmacokinetics of a single dose of RO5185426 and the efficacy and safety of continuous administration in patients with BRAF V600E mutation-positive metastatic melanoma. Patients will be randomized to receive in a crossover design single oral doses of RO5185426 with or without food, with a 10-day washout period between doses. Following the crossover periods, patients will receive RO5185426 orally twice daily on a continuous basis until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically confirmed metastatic melanoma (Stage IV, American Joint Committee on Cancer)
* Positive BRAF V600E mutation result determined by Cobas 4800 BRAF V600 Mutation Test
* Previously treated patients must have failed at least one prior treatment regimen; if patients have received prior systemic treatments for metastatic melanoma, the time elapsed from previous therapy must be >/= 28 days; patients must have recovered fully from toxicities of all prior therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Evaluable disease (measurable for disease progression according to RECIST criteria)
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Active CNS lesions
* History of or known spinal cord compression or carcinomatous meningitis
* Anticipated or ongoing administration of anti-cancer therapies other than those administered in this study
* Previous malignancy within the past 5 years except for basal or squamous cell carcinoma of the skin, melanoma in-situ and carcinoma in-situ of the cervix
* Previous treatment with BRAF inhibitor (sorafenib allowed) or MEK inhibitor
* Refractory nausea or vomiting, malabsorption, external biliary shunt, or history of any type of gastrointestinal surgery that would preclude adequate absorption of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (10):
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lebanon, New Hampshire
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas

REFERENCES:
- [Derived] Frederick DT, Salas Fragomeni RA, Schalck A, Ferreiro-Neira I, Hoff T, Cooper ZA, Haq R, Panka DJ, Kwong LN, Davies MA, Cusack JC, Flaherty KT, Fisher DE, Mier JW, Wargo JA, Sullivan RJ. Clinical profiling of BCL-2 family members in the setting of BRAF inhibition offers a rationale for targeting de novo resistance using BH3 mimetics. PLoS One. 2014 Jul 1;9(7):e101286. doi: 10.1371/journal.pone.0101286. eCollection 2014. PMID 24983357

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib (RO5185426): Fasted Then Fed: Single oral dose of vemurafenib tablet at 960 milligrams (mg) on Day 1 was administered to participants in fasted condition (Period A [Day 1 to Day 10]) followed by single oral dose of vemurafenib tablet at 960 mg on Day 1 in fed condition (Period B [Day 11 to Day 20]). A washout period of 10 days was maintained between Period A and B.
- Vemurafenib (RO5185426): Fed Then Fasted: Single oral dose of vemurafenib tablet at 960 mg on Day 1 was administered to participants in fed condition (Period A [Day 1 to Day 10]) followed by single oral dose of vemurafenib tablet at 960 mg on Day 1 in fasted condition Period B [Day 11 to Day 20]). A washout period of 10 days was maintained between Period A and B.
- Vemurafenib (RO5185426): Participants received vemurafenib tablet at 960 mg orally twice daily in 21-day cycles starting from Day 21 until disease progression, unacceptable toxicity, or consent withdrawal (Period C).
Period: Period A
Arm/Group | Vemurafenib (RO5185426): Fasted Then Fed | Vemurafenib (RO5185426): Fed Then Fasted | Vemurafenib (RO5185426)
Started | 8 | 8 | 0
Completed | 8 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Period B
Arm/Group | Vemurafenib (RO5185426): Fasted Then Fed | Vemurafenib (RO5185426): Fed Then Fasted | Vemurafenib (RO5185426)
Started | 8 | 8 | 0
Completed | 8 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Period C
Arm/Group | Vemurafenib (RO5185426): Fasted Then Fed | Vemurafenib (RO5185426): Fed Then Fasted | Vemurafenib (RO5185426)
Started | 0 | 0 | 16
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 14
Not completed — Disease Progression | 0 | 0 | 4
Not completed — Death | 0 | 0 | 2
Not completed — Follow-up for survival status | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of vemurafenib.
Groups:
- All Participants: Included all participants who received single oral dose of vemurafenib tablet at 960 mg in fasted condition first and fed condition first in Period A and Period B and twice daily dose of vemurafenib tablet at 960 mg in Period C.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.31)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC [0-inf]) in the Fasted and Fed States
Description: Pharmacokinetic (PK) analyses was performed after the completion of Period A and Period B of this study for all participants.
Time Frame: Period A: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16 hours (h) post-dose (pd) on Day 1; 24, 36, 48, 72, 96, 144, 192, and 240 h pd and Period B: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16 h pd on Day 11; 24, 36, 48, 72, 96, 144, 192, and 240 h pd
Population: PK analysis population included participants who received both single doses of vemurafenib in Periods A and B without protocol violation and provided adequate PK assessments to calculate important PK parameters. Here "number of participants analyzed"=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms*hour per milliliter (µg*h/mL)
Groups:
- Vemurafenib (RO5185426): Fasted: Single oral dose of vemurafenib tablet at 960 mg on Day 1 was administered to participants in fasted condition, in any intervention periods (Period A or B).
- Vemurafenib (RO5185426): Fed: Single oral dose of vemurafenib tablet at 960 mg on Day 1 was administered to participants in fed condition, in any intervention periods (Period A or B).
Arm/Group | Vemurafenib (RO5185426): Fasted | Vemurafenib (RO5185426): Fed
Number analyzed (Participants) | 16 | 15
micrograms*hour per milliliter (µg*h/mL) | 115 (110) | 351 (189)
Statistical Analysis 1: Comparison: Vemurafenib (RO5185426): Fasted vs Vemurafenib (RO5185426): Fed; The point estimate and 90 percent (%) confidence interval (CI) of vemurafenib plasma AUC geometric means ratios of the Fed to Fasted conditions following an oral administration of a single dose of 960 mg vemurafenib were analyzed; Test type: Superiority or Other; Ratio of Geometric Mean = 4.64, 90% CI 2-sided [2.83 to 7.60]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Sample With Last Measurable Concentration (AUC[0-last]) in the Fasted and Fed States
Description: PK analyses was performed after the completion of Period A and Period B of this study for all participants.
Time Frame: Period A: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16 h pd on Day 1; 24, 36, 48, 72, 96, 144, 192, and 240 h pd and Period B: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16 h pd on Day 11; 24, 36, 48, 72, 96, 144, 192, and 240 h pd
Population: PK analysis population. Here "number of participants analyzed"=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Vemurafenib (RO5185426): Fasted | Vemurafenib (RO5185426): Fed
Number analyzed (Participants) | 15 | 14
µg*h/mL | 94.3 (81.8) | 320 (158)
Statistical Analysis 1: Comparison: Vemurafenib (RO5185426): Fasted vs Vemurafenib (RO5185426): Fed; The point estimate and 90% CI of vemurafenib plasma AUC geometric means ratios of the Fed to Fasted conditions following an oral administration of a single dose of 960 mg vemurafenib were analyzed; Test type: Superiority or Other; Ratio of Geometric Mean = 5.05, 90% CI 2-sided [2.99 to 8.55]

3. Primary Outcome: Maximal Observed Plasma Concentration (Cmax) in the Fasted and Fed States
Description: PK analyses was performed after the completion of Period A and Period B of this study for all participants.
Time Frame: as for outcome 2
Population: PK analysis population.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Vemurafenib (RO5185426): Fasted | Vemurafenib (RO5185426): Fed
Number analyzed (Participants) | 16 | 16
µg/mL | 3.48 (2.02) | 7.38 (1.98)
Statistical Analysis 1: Comparison: Vemurafenib (RO5185426): Fasted vs Vemurafenib (RO5185426): Fed; The point estimate and 90% CI of vemurafenib plasma Cmax geometric means ratios of the Fed to Fasted conditions following an oral administration of a single dose of 960 mg vemurafenib were analyzed; Test type: Superiority or Other; Ratio of Geometric Mean = 2.45, 90% CI 2-sided [1.81 to 3.32]

4. Primary Outcome: Minimum Observed (Trough) Plasma Concentration (Cmin) in the Fasted and Fed States
Description: Single dose Pre-dose concentration is referred as Cmin here. PK analyses was performed after the completion of Period A and Period B of this study for all participants.
Time Frame: Pre-dose on Periods A and B
Population: PK analysis population.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Vemurafenib (RO5185426): Fasted | Vemurafenib (RO5185426): Fed
Number analyzed (Participants) | 16 | 16
µg/mL | NA (NA) — Since the study was a single-dose study, Cmin was not reached. | NA (NA) — Since the study was a single-dose study, Cmin was not reached.

5. Primary Outcome: Time to Reach Maximal Plasma Concentration (Tmax) in the Fasted and Fed States
Description: PK analyses was performed after the completion of Period A and Period B of this study for all participants.
Time Frame: as for outcome 2
Population: PK analysis population.
Measure: Median (Full Range); unit: hour
Arm/Group | Vemurafenib (RO5185426): Fasted | Vemurafenib (RO5185426): Fed
Number analyzed (Participants) | 16 | 16
hour | 4 [2 to 12.58] | 7.51 [5 to 16]

6. Primary Outcome: Terminal Elimination Half-Life (t1/2) in the Fasted and Fed States
Description: T1/2 is the time required for the concentration of the drug to reach half of its original value. PK analyses was performed after the completion of Period A and Period B of this study for all participants.
Time Frame: as for outcome 2
Population: PK analysis population. Here "number of participants analyzed"=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Vemurafenib (RO5185426): Fasted | Vemurafenib (RO5185426): Fed
Number analyzed (Participants) | 16 | 15
hour | 24.6 (17.2) | 26.0 (17.1)

7. Primary Outcome: Apparent First-order Terminal Elimination Rate Constant (Kel) in the Fasted and Fed States
Description: Apparent first-order terminal elimination rate constant (kel), was calculated as the negative slope of the linear regression of the terminal phase in plasma vemurafenib concentration-time profile using specific appropriate time points. PK analyses was performed after the completion of Period A and Period B of this study for all participants.
Time Frame: as for outcome 2
Population: PK analysis population. Here "number of participants analyzed"=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Vemurafenib (RO5185426): Fasted | Vemurafenib (RO5185426): Fed
Number analyzed (Participants) | 15 | 14
1/h | 0.04 (0.03) | 0.04 (0.02)

8. Secondary Outcome: Percentage of Participants With Best Objective Response (BOR) as Complete Response (CR) or Partial Response (PR)
Description: BOR was defined as the best objective response assessed by investigator during the treatment period according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. BOR was the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation. It is defined as the number of participants whose best objective response was complete response (CR) or partial response (PR) divided by the total number of efficacy evaluable participants. CR: disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes (whether target or non-target) were non-pathological in size (less than [<] 10 millimeter [mm] short axis). PR: at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From Baseline then Day 1 of Cycle 3 and 5 (21-day cycle) at Period C thereafter every 2 cycles until Cycle 12 followed by every 4 cycles from Cycle 13 until disease progression or death (Up to Week 124)
Population: Intent-to-treat (ITT) population included participants with measurable disease who received at least 1 dose of vemurafenib. Here "number of participants analyzed"=participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib (RO5185426)
Number analyzed (Participants) | 14
percentage of participants | 64.3 [35.1 to 87.2]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time, in months, from the date of the first study drug to the date of death, regardless of the cause of death.
Time Frame: From Baseline then Day 1 of Cycle 3 and 5 (21-day cycle) at Period C thereafter every 2 cycles until Cycle 12 followed by every 4 cycles from Cycle 13 until death (Up to Week 124)
Population: Data for OS was not collected as there was a change in planned analysis, not to collect the data.
Arm/Group | Vemurafenib (RO5185426)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose (Week 114)
Groups:
- Vemurafenib (RO5185426): Fasted: Single oral dose of vemurafenib tablet at 960 milligram (mg) on Day 1 was administered to participants in fasted condition, in any intervention periods (Period A or B).
- Vemurafenib (RO5185426): Fed: Single oral dose of vemurafenib tablet at 960 milligram (mg) on Day 1 was administered to participants in fed condition, in any intervention periods (Period A or B).
Arm/Group | Vemurafenib (RO5185426): Fasted | Vemurafenib (RO5185426): Fed | Vemurafenib (RO5185426)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 9/16
Other Adverse Events (participants affected / at risk) | 3/16 | 5/16 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (RO5185426): Fasted (N=16) | Vemurafenib (RO5185426): Fed (N=16) | Vemurafenib (RO5185426) (N=16)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 5
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (RO5185426): Fasted (N=16) | Vemurafenib (RO5185426): Fed (N=16) | Vemurafenib (RO5185426) (N=16)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 2
Blepharitis (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 6
Eye irritation (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Ocular rosacea (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Abdominal distention (Gastrointestinal disorders) | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 5
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 10
Influenza like illness (General disorders) | 0 | 0 | 3
Oedema peripheral (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 2
Breath sounds abnormal (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 1 | 0 | 5
Paraesthesia (Nervous system disorders) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Claustrophobia (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne Conglobata (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 12
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 3
Hypotension (Vascular disorders) | 1 | 1 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1
Dyspnoea Paroxysmal Nocturna (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Results for OS was not reported due to change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.